CLINICAL TRIAL: NCT06633939
Title: The Okla Achokma Project
Acronym: Okla Achokma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Mississippi (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jennifer Lemacks, Associate Dean for Research, University of Southern Mississippi
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 22-880-08; 1R56HL164335-01A1 (NIH)
Record Dates: First submitted 2024-09-26; First posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-09

CONDITIONS: Healthy; Diet; Physical Activity
MeSH Terms: conditions — Motor Activity | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Move & Eat 2 Live (Other): 5, 1-hour sessions with an education and motivational component and focused on nutrition, physical activity and healthy weight.
  Interventions: Behavioral: Behavioral Treatment

INTERVENTIONS:
Behavioral: Behavioral Treatment — The theoretical framework for the Move & Eat 2 Live intervention is guided by the health belief model (HBM), socioecological model (SEM) and motivational interviewing (MI) approach. Tailoring to the target community will include a standard cultural adaptation that will replace curriculum content and examples with Native American relevant foods, physical activities, and representation in materials. For this study, the intervention will be piloted in the target population and will include the first 5 sessions of the original 12-session program.

SUMMARY:
Deep South Native Americans disparately suffer from diabetes, hypertension, and obesity with only 5-10% of Native Americans living past age 65 compared to 15-17% of Whites. Standard lifestyle interventions to improve diet and physical activity behaviors have shown improvement in weight and other cardiometabolic outcomes among Native Americans. The impact of lifestyle interventions on preventable chronic diseases among Native Americans is limited by the exclusion of a multi-level approach with cultural and social enhancements that address the spiritual and social domains of physical health. Therefore, there is an urgent need to determine how spiritual and social domains of health at individual and family levels may advance lifestyle management interventions.

DETAILED DESCRIPTION:
The overall objective for this study is to determine the effectiveness of a more holistic intervention targeting the individual and family levels to enhance health outcomes and program engagement among Native Americans in the Deep South compared to standard approaches. Our central hypothesis is that the integration of spiritual and social domains of health into the standard lifestyle intervention approach will significantly improve attendance, retention, and cardiometabolic profiles of Deep South Native Americans. This hypothesis is supported by our own preliminary data that health behaviors of Deep South Native Americans are fostered by family support and hindered by fatalistic attitudes. The rationale that underlies the proposed research is that demonstration of the feasibility and effectiveness of an intervention that integrates spiritual and social domains will provide new opportunities for its continued development as a strategy to improve disease management/prevention best practices in Deep South Native Americans.

The specific aims for the study are to develop a conceptual model to define spiritual factors and spiritually- and socially-enhanced intervention components that could advance lifestyle management interventions among Native Americans in the Deep South and to determine feasibility of lifestyle intervention components and study instruments among Native Americans in the Deep South. The plan is to to pilot recruitment methods, standard lifestyle intervention components, and implementation protocol and procedures to assess acceptability, optimize population engagement, and improve fidelity of delivery.

ELIGIBILITY:
Inclusion Criteria:

* men or women who self-identify as Native American
* current resident of the Mississippi study site
* at least 18 years of age or older at the time of enrollment
* BMI ≥ 24kg/m2.

Exclusion Criteria:

* individuals with complicated or contraindicated disease diagnosis (i.e., kidney failure or insulin dependent type 2 diabetes) or who are pregnant or within six weeks postpartum

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2024-05-30 (Actual); Primary Completion 2024-08-06 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Program engagement | From first intervention session to the final (5th) intervention session at 10 weeks
  Program engagement will be measured by session attendance and program retention. Session attendance will be captured by the percentage of participants that attend each session. Retention will be examined based on three intervals. Interest retention will include the number of participants who completed the interest form versus those who expressed interest but did not complete the interest form, enrollment retention will include the number of participants who enrolled versus expressed interest but did not enroll, baseline retention will include number of participants who completed baseline data collection versus those who enrolled but did not complete baseline data collection.
Implementation fidelity | from first intervention session to the final (5th) intervention session at 10 weeks
  To examine implementation fidelity, the initial four sessions will be randomly selected for in vivo observation by the primary investigator, co-investigators, and/or research staff. The assessment will be guided by a checklist that includes session information (time, place, session length, etc.), session components, and allows for account of session deviations, etc.

SECONDARY OUTCOMES:
High Density Lipoprotein Cholesterol | at enrollment
  Lipid panel will be measured including cholesterol and High Density Lipoprotein Cholesterol using a portable analyzer and will require a small blood sample from a simple fingerstick.
Health-related quality of life | at enrollment
  A 12-Item Short-Form Health Survey will be used to investigate individual's views about their health. This information will help keep track of how someone feels and how well they are able to do their usual activities.
  Ware, J. E., Kosinski, M., & Keller, S. D. (1996). A 12-Item Short-Form Health Survey: Construction of Scales and Preliminary Tests of Reliability and Validity. Medical Care, 34(3), 220-233. http://www.jstor.org/stable/3766749
Blood Pressure | at enrollment
  systolic and diastolic blood pressure measured in millimeters of mercury (mmHg)
Self-Efficacy | at enrollment
  Validated self-efficacy questionnaire to measure diet and exercise behaviors. Sallis, J.F., Pinski, R.B., Grossman, R.M., Patterson,T.L., and Nader, P.R. (1988). The development of self-efficacy scales for health-related diet and exercise behaviors. Health Education Research, 3, 283-292.
Spirituality | at enrollment
  Holistic assessment instrument focusing on beliefs, intuitions, lifestyle choices, practices, and rituals that represent the human spiritual dimension.
  https://journals.sagepub.com/doi/pdf/10.1177/0898010105276180
Disease Prevention Fatalism | at enrollment
  Validated questionnaire to measure beliefs related to death and disease. Disease Prevention Fatalism: https://pubmed.ncbi.nlm.nih.gov/19908102/
Dietary Intake | at enrollment
  DSQ Dietary Screener Questionnaires (DSQ) in the NHANES 2009-10: DSQ https://epi.grants.cancer.gov/nhanes/dietscreen/questionnaires.html#paper
Physcial Activity | at enrollment
  Validated International Physical Activity Questionnaire, short form. IPAQ_English_telephone_short.pdf. (n.d.). https://www.google.com/url?sa=t&source=web&rct=j&opi=89978449&url=https://osf.io/6yfjf/&ved=2ahUKEwiKn5S0l_OIAxXyG9AFHVV0OlsQFnoECBoQAQ&usg=AOvVaw1JvoOLn0pQMye2UUBQt_DX

OTHER OUTCOMES:
Girth circumference | at enrollment
  Waist, abdomen, and hip circumferences will be measured with a plastic, non-flexible, circumference measuring tape as the participant exhales.
Weight | at enrollment
  Measured in lightweight clothing without shoes to the nearest 0.1kg/%.
Height | enrollment
  Height will be measured without shoes using a stadiometer in ft and inches.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Lemacks, PhD, Principal Investigator — The University of Southern Mississippi
Locations (1):
- The University of Southern Mississippi, Hattiesburg, Mississippi, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lemacks JL, James RE, Abbott L, Choi H, Parker A, Bryant A, Ralston PA, Rigsby AG, Gilner P. The Church Bridge Project: An Academic-Community Perspective of a Church-Based Weight Management Pilot Intervention among Young Adult African Americans. Prog Community Health Partnersh. 2018;12(1S):23-34. doi: 10.1353/cpr.2018.0018. PMID 29755046
- [Background] Abbott L, Lemacks J, Greer T. Development and Evaluation of a Measure for Social Support Provided by Friends during Lifestyle Management Programs. Healthcare (Basel). 2022 May 13;10(5):901. doi: 10.3390/healthcare10050901. PMID 35628038